CLINICAL TRIAL: NCT05790772
Title: Biochemical Changes in Blood Plasma After Intense Physical Exercise of Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Touro University Nevada (Other)
Responsible Party: Principal Investigator, Derek Tai, Principal Investigator, Touro University Nevada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TUNIRB000225
Record Dates: First submitted 2023-03-06; First posted 2023-03-30 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Hormone Disturbance; Endorphin Changes
MeSH Terms: conditions — Endocrine System Diseases

STUDY DESIGN:
Intervention Model Description: 20 Male and Female Athletes Aged 18-65
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vigorous Exercise (Experimental): 50 Minutes of running on a treadmill
  Interventions: Behavioral: Vigorous Exercise

INTERVENTIONS:
Behavioral: Vigorous Exercise — 50 minutes of running on a treadmill

SUMMARY:
This study will recruit 20 male and female athletes of endurance training background. They will participate in 50 minutes of vigorous activity on a treadmill with 3 blood draws (before exercising, 50 minutes into exercising, and 30 minutes after completion of exercising). After collection of the blood samples, the results will be analyzed for extracellular vesicles and biochemical changes within said extracellular vesicles.

DETAILED DESCRIPTION:
This study will recruit participants from the Touro University Nevada student body by placing flyers around campus and including announcements on the TUN screens. Program faculty will be encouraged to promote the study to their students through March.

20 male and female athletes who currently participate in regular endurance training will be recruited for the study. We will use men because the hormonal responses to exercise vary between men and women and is blunted at different points during the reproductive cycle. Participants recruited into the study will be normal weight (BMI or waist-to-hip ratio), and a history of regular participation in endurance training (see flyer). Participants will not have been diagnosed or treated for any psychiatric conditions, lower extremity or low back injury and will not have regularly taken any prescription medications within the past year.

Participants will be consented into the study, scheduled, and given pre-participation instructions one week prior to the event. They will not take over-the-counter medications or supplements within one week of the trial, have no alcohol within 72 hours and no caffeine or nicotine within four hours, and no food within two hours of the protocol. Participants may drink water ad libitum prior to the trial.

Upon arriving the day of the trial, participants will be screened by urinalysis for drug use. They will complete a survey based on the International Physical Activity Questionnaire which will be used to classify their history of physical activity. They will complete a pre-activity screen of their current emotional state using a set of Visual Analog Scales (VAS).

On the day of the trial, participants will provide a urine sample for urinalysis. They will complete an electronic survey on their cell phone and will complete a paper survey including a set of visual analog scales. A butterfly needle will be inserted into their arm of choice which will allow the four small (5 ml) blood samples to be drawn throughout the activity. The first sample will be drawn immediately upon inserting the needle with subsequent draws performed at 50-minutes of physical activity, and the final draw 30-minutes after the activity ends. They will wear a heart monitor that will be used to monitor exercise intensity throughout the exercise protocol.

Participants will complete an exercise protocol that includes 50 minutes of vigorous activity on a treadmill. They will be instructed to perform a 5-minute warm up and then begin running at a rate and treadmill elevation that ensures that they are working at 76-96% of their age-adjusted maximum heart rate. An attendant will monitor their heart rate throughout the protocol to ensure compliance. The participant will continue to exercise while blood is drawn at 50-minutes of activity.

A butterfly needle will be inserted into the arm of their choice. A baseline sample of 5 ml of blood will be drawn immediately with subsequent 5 ml samples drawn at 25- and 50-minutes into the exercise protocol. A final 5 ml sample will be drawn at 30 minutes after completion of the protocol. The butterfly needle will be removed immediately after the final blood draw.

The endorphin response has been documented at 70% of age-adjusted maximum heart rate and increases linearly after that. A heart monitor will be worn throughout the trial to monitor exercise intensity which will be determined based on the ACSM guidelines for vigorous exercise, 76-96% of the participant's age-adjusted maximum heart rate (AAMHR). Participants will be instructed to perform a 5-minute warm up and then begin running. A monitor will ensure that the participant maintains the target intensity throughout the activity.

After completing the physical activity, participants will be offered healthy snacks while they walk, sit, or lie down anywhere within the lab. They will complete the second set of VAS ratings of emotional state that will be used to differentiate runners who experience "runner's high" from those who do not. The final 5 ml of blood will be drawn 30 minutes after completion of the exercise protocol after which the participant will take off the heart monitor and leave the lab.

After collection of the blood samples, the results will be separated into blood plasma. The blood plasma will be analyzed for extracellular vesicles and quantitative biochemical changes within said extracellular vesicles.

ELIGIBILITY:
Inclusion Criteria:

* Has reportedly experienced "runner's high" during vigorous exercise.

Exclusion Criteria:

* Has not reportedly experienced "runner's high" during vigorous exercise.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-07-23 (Actual)

PRIMARY OUTCOMES:
Biochemical Changes in Blood Plasma | 0 minutes into exercising
  Endorphin expression (AU arbitrary unit) in Extracellular Vesicles within Blood Plasma via Western Blot
Biochemical Changes in Blood Plasma | 50 minutes into exercising
  Endorphin expression (AU arbitrary unit) in Extracellular Vesicles within Blood Plasma via Western Blot
Biochemical Changes in Blood Plasma | 30 minutes after completion of exercising
  Endorphin expression (AU arbitrary unit) in Extracellular Vesicles within Blood Plasma via Western Blot

CONTACTS AND LOCATIONS:
Locations (1):
- Touro University Nevada, Henderson, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be made anonymous to protect their identity as data analysis begins.